

# STATISTICAL ANALYSIS PLAN

The TRANQUILITY Trial: A Multi-Center Randomized, Double-Masked, Parallel Design, Vehicle-Controlled Phase 2/3 Clinical Trial to Assess the Efficacy and Safety of 0.25% Reproxalap Ophthalmic Solution Compared to Vehicle in Subjects with Dry Eye Disease

Sponsor: Aldeyra Therapeutics, Inc.

Protocol Number: ADX-102-DED-019

Author:

Date: 17-NOV-2021

Version: 2.0



The TRANQUILITY Trial: A Multi-Center Randomized, Double-Masked, Parallel Design, Vehicle-Controlled Phase 2/3 Clinical Trial to Assess the Efficacy and Safety of 0.25% Reproxalap Ophthalmic Solution Compared to Vehicle in Subjects with Dry Eye Disease

Protocol Number: ADX-102-DED-019

SAP Version: 2.0

SAP Date: 17-NOV-2021

### **Statistical Analysis Plan Approval**















### **Document History**

SignNow E-Signature Audit Log All dates expressed in MM/DD/YYYY (US)

**Document name:** Aldeyra ADX-102-DED-019 Statistical Analysis Plan V2.0 17-NOV-2021

**Document created:** 11/17/2021 22:20:14

Document pages: 41

**Document ID:** 32f5fbfe725245dca5b1a6008fa3f33e31893ae2

**Document Sent:** 11/17/2021 22:20:48 UTC

**Document Status:** Signed

11/17/2021 23:39:40UTC











### **Table of Contents**

| 1. | | Introduction | g |
|---|---|---|---|
| 2. | | Study Objectives | 9 |
| 3. | | Study Endpoints | 9 |
| | 3.1 | Primary Endpoints | 9 |
| | 3.2 | Secondary Variables | 9 |
| | 3.3 | Exploratory Variables | 9 |
| | 3.4 | Safety Variables | . 10 |
| | 3.5 | Statistical Hypotheses | . 10 |
| | 3.6 | Estimands | . 10 |
| 4. | | Study Design and Procedures | .11 |
| | 4.1 | General Study Design | . 11 |
| | 4.2 | Schedule of Visits and Assessments | . 12 |
| 5. | | Study Treatments | .13 |
| | 5.1 | Method of Assigning Subjects to Treatment Groups | . 13 |
| | 5.2 | Masking and Unmasking | . 13 |
| 6. | | Sample Size and Power Considerations | .13 |
| 7. | | Data Preparation | .14 |
| | 7.1 | Input Data | . 14 |
| | 7.2 | Output Data | . 14 |
| 8. | | Analysis Populations | . 15 |
| | 8.1 | Intent-to-Treat. | . 15 |
| | 8.2 | Initial Cohort | . 15 |
| | 8.3 | Per Protocol | . 15 |
| | 8.4 | Safety | . 15 |
| 9. | | General Statistical Considerations | .15 |
| | 9.1 | Unit of Analysis | . 15 |
| | 9.2 | Missing or Inconclusive Data Handling | . 15 |
| | 9.3 | Definition of Baseline | . 16 |
| | 9.4 | Data Analysis Conventions | . 16 |
| | 9.5 | Adjustments for Multiplicity | . 17 |
| 10 | ). | Disposition of Subjects | .17 |
| 11 | | Demographic, Previous Participation in Reproxalap Trials, and Pretreatment Variables | .18 |
| | 11.1 | Demographic Variables | .18 |
| | 11.2 | Previous Participation in Reproxalap Trials | .18 |
| | 11.3 | Pretreatment Variables | . 19 |
| 12 | 2. | Medical History and Concomitant Medications | .19 |



| 12.1 Med | dical History | 19 |
|---|---|---|
| 12.2 Con | ncomitant Medications and Procedures | 19 |
| 13. Dos | sing Compliance and Treatment Exposure | 20 |
| 13.1 Dos | sing Compliance | 20 |
| 13.2 Trea | atment Exposure | 20 |
| 14. Effic | cacy Analyses | 20 |
| 14.1 Prim | nary Analysis | 21 |
| 14.1.1<br>14.1<br>14.1<br>14.1 | .1.1 Mixed Model Repeated Measures .1.2 Mixed Model Repeated Measures | 22<br>22 |
| 14.2 Sec | condary Analyses | 23 |
| 14.2.1 | Overall Mean Change from Baseline of Eye Dryness Score (VAS) | 23 |
| 14.2.2 | <u> </u> | |
| 14.2.3 | | 24 |
| | oloratory Analyses | 25 |
| 14.3.1 | Eye Dryness Score from the Visual Analog Scale | |
| 14.3.2 | Ocular Discomfort Scale (Ora Calibra® Scale) | |
| 14.3.3<br>14.3<br>14.3 | 3.3.1 Ocular Discomfort & 4-Symptom Questionnaire (Ora Calibra® Ścale) | 26 |
| 14.3 | 3cale) | |
| 14.3.4<br>14.3 | - , | |
| 14.3 | 3.4.2 Conjunctival Allergen Challenge Ocular Itching Scale (Ora Calibra <sup>®</sup> Scale | e) |
| 14.3.5<br>27 | Conjunctival Redness | |
| 14.3.6 | Tear Reactive Aldehyde Species | 27 |
| 14.3.7 | Conjunctival Redness (Ora Calibra® Scale) | |
| 14.3.8 | Eye Dryness (VAS) | 28 |
| 14.3.9<br>28 | Ocular Discomfort Scale (Ora Calibra® Scale) | |
| 15. Effic | cacy Analyses of the Initial Cohort | 28 |
| 16. Sun | mmary of Efficacy Analyses | 29 |
| 17. Safe | ety Analyses | 29 |
| 17.1 Adv | verse Events | 29 |



| 17 | 7.1.1 | Severity | 30 |
|---|---|---|---|
| 17 | 7.1.2 | Relationship to Study Procedures | .31 |
| 17 | 7.1.3 | Expectedness | .31 |
| 17 | 7.1.4 | Serious Adverse Events | .32 |
| 17.2 | 2 Visual <i>i</i> | Acuity (Early Treatment Diabetic Retinopathy Study) | .32 |
| 17.3 | Slit-Lar | np Biomicroscopy | .33 |
| 17.4 | Dilated | Fundoscopy Examination | 33 |
| 17.5 | Intraoc | ular Pressure (IOP) | .33 |
| 18. | Change | es from Protocol-Stated Analyses | .33 |
| 19. | Refere | nces | .33 |
| 20. | Revisio | n History | .33 |
| 21. | Tables | | .34 |
| 22. | Listings | 3 | 39 |



### **List of Abbreviations**

| ADaM | Analysis Data Model |
|--------|-----------------------------------------------|
| AE | Adverse Event |
| ANCOVA | Analysis of Covariance |
| ATC | Anatomical Therapeutic Chemical |
| CAC | Conjunctival Allergen Challenge |
| CAE® | Controlled Adverse Environment® |
| CI | Confidence Interval |
| CS | Clinically Significant |
| DED | Dry Eye Disease |
| eCRF | Electronic Case Report Form |
| EDC | Electronic Data Capture |
| ETDRS | Early Treatment of Diabetic Retinopathy Study |
| ICH | International Conference on Harmonisation |
| IOP | Intraocular Pressure |
| ITT | Intent-to-Treat |
| IWRS | Interactive Web Response System |
| logMAR | Logarithm of the Minimum Angle of Resolution |
| LS | Least Squares |
| MAR | Missing at Random |
| MCMC | Markov Chain Monte Carlo |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MMRM | Mixed Model Repeated Measures |
| MNAR | Missing Not at Random |
| NCS | Not Clinically Significant |
| OD | Oculus dexter (Right Eye) |
| OS | Oculus sinister (Left Eye) |
| PDF | Portable Document Format |
| PMM | Pattern Mixture Model |
| PP | Per Protocol |
| PT | Preferred Term |
| RASP | Reactive Aldehyde Species |
| RDC | Remote Data Capture |
| RTF | Rich Text Format |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SDC | Statistics & Data Corporation |
| SDTM | Study Data Tabulation Model |
| SE | Standard Error |
| SOC | System Organ Class |
| TEAE | Treatment-Emergent Adverse Event |
| TMF | Trial Master File |
| VAS | Visual Analog Scale |



| MILIOD | W |
|-----------|-------------------------------------------|
| WHODrug | World Health Organization Drug Dictionary |
| vviiobiag | World Hoalth Organization Brag Blottonary |



#### 1. Introduction

The purpose of this statistical analysis plan (SAP) is to describe the planned analyses and reporting for protocol ADX-102-DED-019, Amendment 3.0, dated 5-NOV-2021.

This SAP is being written with due consideration of the recommendations outlined in the most recent International Conference on Harmonisation (ICH) E9 Guideline entitled Guidance for Industry: Statistical Principles for Clinical Trials, E9(R1) Statistical Principles for Clinical Trials: Addendum: Estimands and Sensitivity Analysis in Clinical Trials, and the most recent ICH E3 Guideline entitled Guidance for Industry: Structure and Content of Clinical Study Reports.

This SAP describes the data that will be analyzed and the subject characteristics, efficacy, and safety assessments that will be evaluated. This SAP provides details of the specific statistical methods that will be used. The statistical analysis methods presented in this document will supersede the statistical analysis methods described in the clinical protocol. If additional analyses are required to supplement the planned analyses described in this SAP, they may be completed and will be identified in the clinical study report.

#### 2. Study Objectives

To evaluate the efficacy of reproxalap, as assessed by conjunctival redness, tear reactive aldehyde species (RASP) levels, Schirmer's Test, and symptoms after dosing to the Controlled Adverse Environment® (CAE®) in subjects with dry eye disease (DED).

### 3. Study Endpoints

#### 3.1 Primary Endpoints

The primary efficacy variable is the following:

Conjunctival redness

### 3.2 Secondary Variables

The secondary efficacy variables are the following:

- Visual analog scale (VAS) eye dryness score
- Ora Calibra<sup>®</sup> Ocular Discomfort Scale



Schirmer's Test

### 3.3 Exploratory Variables

The exploratory efficacy variables are the following:

- VAS eye dryness score
- Ora Calibra<sup>®</sup> Ocular Discomfort Scale



| Ocular Discomfort & | 4-Symptom Questionnaire |
|---|---|
| Ora Calibra® Canius | etivel Allegge Chellenge Couley Itching Coole |
| Ora Calibra Conjun | ctival Allergen Challenge Ocular Itching Scale |
| Change in tear RASI | Pievels |
| Conjunctival redness | |
| | s, Ora Calibra <sup>®</sup> Ocular Discomfort Scale, and VAS dryness score |
| o Conjunctival realises | , Ora Gallista Godial Discontinist Godie, and VAG dryficos Soore |
| 3.4 Safety Variables | |
| The safety variables include | the following: |
| <ul> <li>Visual acuity</li> </ul> | |
| Slit-lamp evaluation | |
| Adverse event (AE) | query |
| Intraocular Pressure | |
| Dilated fundoscopy | |
| 3.5 Statistical Hypothe | 202 |
| | be tested comparing reproxalap to vehicle. The null hypothesis |
| must be rejected for the dosi | |
| | ig regimen to elamin emedey. |
| 3.6 Estimands | |
| The primary comparisons in | this trial will be between reproxalap versus vehicle |
| Estimand 1 | |
| • | |





### 4. Study Design and Procedures

### 4.1 General Study Design

Study visits will be referred to in all tables and listings as the expected study day corresponding to the visit to enable reviewers to understand the assessment timing without referring to the protocol visit schedule. Table 1 shows the scheduled study visits, their planned study day (note that there is no Day 0 and that Day 1 corresponds to the day of randomization), and the acceptable visit window for each study visit:

**Table 1. Study Visit Windows** 

| Scheduled Visit | Planned Study Day | Visit Window |
|-----------------|-------------------|--------------|
| Visit 1 | Day -14 | -16/+2 days |
| Visit 2 | Day 1 | N/A |
| Visit 3 | Day 2 | N/A |



# 4.2 Schedule of Visits and Assessments

**Table 2. Schedule of Visits and Assessments** 





### 5. Study Treatments

#### 5.1 Method of Assigning Subjects to Treatment Groups

At Visit 1 (Day -14), each subject who signs the informed consent will be assigned a screening number. All screening numbers will be assigned in strict numerical sequence at each site and no numbers will be skipped or omitted.

At Visit 2 (Day 1), a subject who meets all the eligibility criteria will be randomized in a 1:1 ratio to receive treatment with either 0.25% Reproxalap Ophthalmic Solution or placebo. Subjects will be assigned a randomization number and kit number via paper randomization list for the Initial Cohort and by interactive web response system (IWRS) for the Main Cohort.

The site staff will dispense to the subject the study kit labeled with the corresponding kit number. Both the randomization number and the dispensed study drug kit number will be recorded on the subject's source document and electronic case report form (eCRF).

#### 5.2 Masking and Unmasking

All subjects, investigators, and study personnel involved with the conduct of the study will be masked with regard to treatment assignments. When medically necessary, the investigator may need to determine what treatment arm has been assigned to a subject. When possible (i.e., in non-emergent situations), Ora and/or the study Sponsor should be notified, when possible, before unmasking study drug as described in the following paragraph.

If an investigator identifies a medical need for unmasking the treatment assignment of a subject, he/she should contact Ora and/or the medical monitor prior to unmasking the identity of the IP, if possible. Ora will ask the site to complete and send them the Unmasking Request Form. Ora will notify Aldeyra and jointly will determine if the unmasking request should be granted. They may consult the medical monitor as needed. The result of the request will be documented on the Unmasking Request Form. If approval is granted to unmask a subject, written permission via the Unmasking Request Form will be provided to the investigator. The investigator will unmask the subject via scratch off labels on the kits for the Initial Cohort Only. The investigator will unmask the subject using IWRS for the Main Cohort. The investigator will complete the Unmasking Memo form and include it in the subject's study file and provide a copy for the Trial Master File (TMF). For each unmasked request, the reason, date, signature, and name of the person who unmasked the subject, must be noted in the subject's study file.

Planned unmasking was executed for subjects in the initial cohort for sample size and power calculations.

# 6. Sample Size and Power Considerations





# 7. Data Preparation

#### 7.1 Input Data

Study data will primarily be recorded on the eCRFs supplied by Statistics & Data Corporation (SDC) using is delivered as a single-instance, multitenant and is developed, maintained, and hosted by These data sources are described in detail in data transfer agreements developed between data management and the respective external laboratory or reading center:

- Tear RASP data
- Conjunctival redness photography scores

When all prerequisites for database lock have been met, including availability of all masked external data, the database will be locked. Following database lock, approval will be obtained from the Sponsor to unmask the study. Once the study has been unmasked, unmasked laboratory data will be sent to SDC. Any changes to the database after data have been locked can only be made with the approval of the Sponsor in consultation with SDC.

Final analysis will be carried out after the following have occurred:

- Database lock has occurred, including receipt of all final versions of external vendor data, with written authorization provided by appropriate SDC and Sponsor personnel.
- Protocol deviations have been identified and status defined (major/minor deviations).
- Analysis populations have been determined.
- Randomized treatment codes have been unmasked.

#### 7.2 Output Data

| Data from EDC and external data will be tran | nsferred to SDC Biostatistics and incorporated into sta | ndard |
|---|---|---|
| formats following the | | |
| SDTM will follow the | I and will be implemented using the | |
| | at the time of study | start |
| _ | | |



#### 8. Analysis Populations

#### 8.1 Intent-to-Treat

The Intent-to-Treat (ITT) Population includes all randomized subjects. Subjects in the ITT Population will be analyzed as randomized. Subjects in the initial cohort will not be included in the ITT Population for efficacy analyses.

| ; |
|---|

#### 8.2 Initial Cohort

The Initial Cohort Population includes all randomized subjects in the Initial Cohort. Subjects in the Initial Cohort will be analyzed as randomized.

#### 8.3 Per Protocol

The Per-Protocol (PP) Population includes subjects in the ITT Population who do not have significant protocol deviations and who complete the study. Protocol deviations will be assessed prior to database lock and unmasking. Subjects in the PP Population will be analyzed as treated.

#### 8.4 Safety

The Safety Population includes all randomized subjects who receive at least one dose of investigational product. Subjects in the Safety Population will be analyzed as treated. The Safety Population includes subjects in the initial cohort who receive at least one dose of investigational product.

#### 9. General Statistical Considerations

### 9.1 Unit of Analysis

| Safety endpoints will be analyzed |
|-----------------------------------|

#### 9.2 Missing or Inconclusive Data Handling

Partial/missing start and end dates for AEs and concomitant medications required to flag data as treatmentemergent or concomitant with treatment will be imputed as follows:



| • |
|---|
| Partial/missing end date: |
| • |
| The PP population analysis will also be conducted t |
| assess sensitivity. |
| 9.3 Definition of Baseline |
| Baseline is defined |
| 9.4 Data Analysis Conventions |
| All data analysis will be performed by SDC after the study is completed and the database has been locke |
| and released for unmasking. Statistical programming and analyses will be performed |



| 9.5 Adjustments for Multiplicity |
|---|
| The primary endpoint of the overall mean change from baseline of conjunctival redness |
| 10. Disposition of Subjects |
| Subject disposition will be presented in terms of the numbers and percentages of subjects who were |
| randomized |



| In addition, a listing of all subjects affected by |
|---|
| COVID-19 will be produced. |
| 11. Demographic, Previous Participation in Reproxalap Trials, and Pretreatment Variables |
| 11.1 Demographic Variables |
| The demographic variables collected in this study |
| Age (years) will be summarized, overall and by treatment, using continuous descriptive statistics. |

A subject listing that includes all demographic variables including informed consent will be provided.

### 11.2 Previous Participation in Reproxalap Trials

The number of subjects and percentages of subjects that dosed with randomized study drug in previous Reproxalap trials will be summarized by treatment group and for all subjects in the ITT population.





| Subjec | ts who did not dose under previous Reproxalap studies will be summarized as well. |
|---|---|
| 11.3 | Pretreatment Variables |
| All bas | eline efficacy and safety variables will be summarized |
| | Summaries will be provided of the ITT and |
| Safety | Populations. |
| 12. Me | edical History and Concomitant Medications |
| 12.1 | Medical History |
| Medica | al history will be coded using Medical Dictionary for Regulatory Activities . |
| _ | · |
| Listing | s of medical history will be generated separately for ocular and non-ocular data. |
| 12.2 | Concomitant Medications and Procedures |
| Concomitant medications and procedures will be coded using World Health Organization Drug Dictional | |



| Listings |
|---|
| of concomitant medications will be generated separately for ocular and non-ocular data. |
| 13. Dosing Compliance and Treatment Exposure |
| 13.1 Dosing Compliance |
| Dosing compliance (% compliance) will be assessed |
| A subject listing of dosing compliance will also be produced. |
| 13.2 Treatment Exposure |
| Extent of treatment exposure for subjects |
| . A subject listing of treatment |
| exposure will also be produced. |
| 14. Efficacy Analyses |
| All efficacy analyses described in this section will have SAS code specified in the SAP |



# 14.1 Primary Analysis

| The primary endpoint will be deemed to have been met |
|------------------------------------------------------|
| 14.1.1 PRIMARY ANALYSES METHODS |
| The endpoint of overall mean change from baseline |



| 14.1.1.1 | MIXED MODEL REPEATED MEASURES |
|--------------|---------------------------------|
| Overall mean | change from baseline |
| 14.1.1.2 | MIXED MODEL REPEATED MEASURES |
| 14.1.1.2 | WINED WIODEL NEI EATED WEAGONES |



| 14.1.1.3 ADDITIONAL SENSITIVITY ANALYSES |
|-----------------------------------------------------------------|
| Additional sensitivity analyses will be performed |
| <u> </u> |
| 14.2 Secondary Analyses |
| 14.2.1 OVERALL MEAN CHANGE FROM BASELINE OF EYE DRYNESS SCORE ( |
| Subjects will be |
| Subjects will be |
| - |
| . A subject listing of the eye dryness duri |
| the CAE will be generated. |



| 14.2.2 OVERALL MEAN CHANGE FROM BASELINE OF OCULAR DISCOMFORT SCALE (ORA CALIBRA® SCALE) |
|---|
| Ocular Discomfort will be accessed |
| Ocular Discomfort will be assessed |
| <u>-</u> |
| A subject listing of the Ocular Discomfort |
| Scale during the CAE® will be generated. |
| 14.2.3 UNANESTHETIZED SCHIRMER'S TEST |
| Unanesthetized Schirmer's test will be assessed for each eye. |
| A publicat listing of the |
| A subject listing of the unanesthetized Schirmer's test will be generated. |
| unanesinetized schiinners test wiii be generated. |



# 14.3 Exploratory Analyses

| 14.3.1 EYE DRYNESS SCORE FROM THE VISUAL ANALOG SCAL | E STATE OF THE STA |
|---|---|
| Subjects will be asked to rate eye dryness | |
| of the CAT® will be accompanded | A subject listing of the eye dryness outside |
| of the CAE <sup>®</sup> will be generated. | <u></u> |
| 14.3.2 OCULAR DISCOMFORT SCALE (ORA CALIBRA® SCALE) | |
| Ocular Discomfort Scale will be assessed | |



A subject listing of the Ocular Discomfort Scale outside of the CAE® will be generated. 14.3.3 OCULAR DISCOMFORT & 4-SYMPTOM QUESTIONNAIRE (ORA CALIBRA® SCALE) Ocular Discomfort and dry eye symptoms will be assessed A subject listing of the Ocular Discomfort & 4-Symptom Questionnaire will be generated. OCULAR DISCOMFORT & 4-SYMPTOM QUESTIONNAIRE (ORA CALIBRA® SCALE) Overall mean CFB of each Ocular Discomfort & 4-Symptom Questionnaire A subject listing of the Ocular Discomfort & 4-Symptom Questionnaire will be generated. 14.3.4 CONJUNCTIVAL ALLERGEN CHALLENGE OCULAR ITCHING SCALE (ORA CALIBRA® SCALE) Subjects will rate the severity of their ocular itching symptom CONJUNCTIVAL ALLERGEN CHALLENGE OCULAR ITCHING SCALE (ORA CALIBRA® SCALE) Overall mean CFB of ocular itching



| A subject listing of the Conjunctival A | Allergen |
|---|---|
| Challenge Ocular Itching Scale will be generated. | |
| 14.3.4.2 CONJUNCTIVAL ALLERGEN CHALLENGE OCULAR ITCHING SCALE (ORA CALIBRA® | Scale) |
| Overall mean CFB of ocular itching | |
| <u> </u> | |
| 14.3.5 CONJUNCTIVAL REDNESS (ORA CALIBRA SCALE | |
| Each subject eye at each visit/time point will be assessed | |
| A subject listing of the conjunctival r | redness |
| outside of the CAE® will be generated. | |
| 14.3.6 TEAR REACTIVE ALDEHYDE SPECIES | |
| Tears will be collected | |



| A cubic of lighting of the Acon DACD will |
|-----------------------------------------------------|
| A subject listing of the tear RASP will |
| generated. |
| 14.3.7 CONJUNCTIVAL REDNESS (ORA CALIBRA® SCALE) |
| For conjunctival redness during the CAE® |
| 14.3.8 EYE DRYNESS (VAS) |
| For eye dryness (VAS) |
| 14.3.9 OCULAR DISCOMFORT SCALE (ORA CALIBRA® SCALE) |
| For ocular discomfort |
| 1 of occide disconnect |

### 15. Efficacy Analyses of the Initial Cohort

All efficacy analyses stated in section 14 using the ITT population will be repeated using the Initial Cohort only with the following exceptions:





### 16. Summary of Efficacy Analyses

A summary of all efficacy analyses will be presented.

#### 17. Safety Analyses

All safety analyses will be conducted using the Safety Population using observed data only.

#### **Adverse Events** 17.1

For the purposes of this trial, an AE is defined as any untoward medical event occurring after the subject's signing of the informed consent until they are exited from the trial. An AE can therefore be any unfavorable and unintended sign, symptom, or disease occurring after the subject started the clinical trial, without any judgment about causality. Any pre-existing medical condition that worsens during the trial will also be considered a new AE. Documentation regarding the AE should be made as to the nature, date of onset, end date, severity, relationship to study procedure, expectedness, action(s) taken, seriousness, and outcome of any sign or symptom observed by the investigator or reported by the patient upon indirect questioning.

All AEs will be coded using the MedDRA

Treatment-emergent adverse events (TEAEs) are defined as any event that occurs or worsens on or after the day that randomized study treatment is initiated. Adverse events recorded in the eCRF which began prior to treatment will not be included in the summary tables but will be included in the AE data listings.

An overall summary will be presented that includes the number and percentage of subjects who experienced at least one AEs, ocular AEs, non-ocular AEs, SAEs, AEs by maximal severity, AEs by



relationship to study procedure, AEs leading to treatment discontinuation, and AEs resulting in death by treatment arm for the Safety Population. In addition, overall TEAEs and the number and percentage of subjects who experienced at least one TEAE, ocular TEAEs, non-ocular TEAEs, TE-SAEs, TEAEs by maximal severity, TEAEs by relationship to study procedure, TEAEs leading to treatment discontinuation, and TEAEs resulting in death by treatment arm for the Safety Population.

Separate summaries will be provided for the following categories of AEs:

- Ocular AEs by SOC and PT
- Non-ocular AEs by SOC and PT
- Ocular TEAEs by SOC and PT
- Non-ocular TEAEs by SOC and PT
- Instillation Site Ocular TEAEs by Duration of Time
- Ocular TEAEs by SOC, PT, and maximal severity
- Non-ocular TEAEs by SOC, PT, and maximal severity
- Ocular TEAEs by SOC, PT, and strongest relationship to study procedure
- Non-ocular TEAEs by SOC, PT, and strongest relationship to study procedure
- Ocular TEAEs by SOC, PT, maximal severity, and strongest relationship to study procedure
- Non-ocular TEAEs by SOC, PT, maximal severity, and strongest relationship to study procedure
- TEAEs That Led to Premature Treatment Discontinuation
- SAEs

Adverse Events and TEAEs will be summarized using discrete summary statistics and presented by treatment arm and all subjects for the the Safety Population. If a subject reports the same PT multiple times within the same SOC, that PT will only be reported once within that SOC. As with the PT, if a subject reports multiple conditions within the same SOC, that SOC will only be reported once. In the summaries, SOCs will be listed in ascending alphabetical order. PTs will be listed in order of descending frequency within each SOC for all subjects..

All AEs, ocular AEs, non-ocular AEs, and SAEs will be presented in subject listings.

#### **17.1.1 SEVERITY**

Severity of an AE is defined as a qualitative assessment of the degree of intensity of an AE as determined by the investigator or reported to him/her by the patient/subject. The assessment of severity is made irrespective of relationship to study procedures or seriousness of the event and should be evaluated according to the following scale:



| • |
|---|

Subjects experiencing more than one AE within a given SOC or PT are counted once within that SOC or PT for the maximal severity.

#### 17.1.2 RELATIONSHIP TO STUDY PROCEDURES

The relationship of each AE to the study procedures should be determined by the investigator using these explanations. Decisive factors for the assessment of causal relationship of an AE to the study procedures include, but may not be limited to, temporal relationship between the AE and the procedure, known side effects of the procedure medical history, and/or concomitant medication:

- Definite: When there are good reason and sufficient documentation to demonstrate a direct causal relationship between study procedure and AE;
- Probable: When there are good reasons and sufficient documentation to assume a causal relationship in the sense of plausible, conceivable, likely but not necessarily highly probable.
- Possible: When there is sufficient information to accept the possibility of a causal relationship in the sense of not impossible and not unlikely, although the connection is uncertain or doubtful, for example; due to missing data or insufficient evidence.
- None: When there is sufficient information to accept a lack of a causal relationship, in the sense of impossible and improbable.
- Unclassified: When the causal relationship is not assessable for whatever reason due to insufficient evidence, conflicting data or poor documentation.

Subjects experiencing more than one AE within a given SOC or PT are counted once within that SOC or PT for the maximum relationship.

#### 17.1.3 EXPECTEDNESS

The expectedness of an AE should be determined based upon existing safety information about the study procedures. Therefore, the following definition will be used:

- Unexpected: An AE that is not listed in the safety information available for the study procedure at the specificity or severity that has been observed.
- Expected: An AE that is listed in the safety information available for the study procedure at the specificity and severity that has been observed.
- Not Applicable: Any AE that is unrelated to the study procedure.



#### 17.1.4 SERIOUS ADVERSE EVENTS

An AE is considered serious if, in the view of either the investigator or sponsor, it results in any of the following outcomes:

- Death;
- A life-threatening adverse event;
  - Note: An adverse event is considered "life-threatening" if, in the view of either the
    investigator or sponsor, its occurrence places the patient or subject at immediate risk of
    death. It does not include an adverse event that, had it occurred in a more severe form,
    might have caused death.
- Inpatient hospitalization or prolongation of existing hospitalization;
  - Note: The term "inpatient hospitalization" refers to any inpatient admission (even if less than 24 hours). For chronic or long-term inpatients, inpatient admission includes transfer within the hospital to an acute/intensive care inpatient unit. Inpatient hospitalization does not include: emergency room visits; outpatient/same-day/ambulatory procedures; observation/short stay units; rehabilitation facilities; hospice facilities; nursing homes; or clinical research/phase 1 units.
  - Note: The term "prolongation of existing hospitalization" refers to any extension of an inpatient hospitalization beyond the stay anticipated or required for the reason for the initial admission as determined by the investigator or treating physician.
- A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions;
  - Note: A serious adverse event specifically related to visual threat would be interpreted as any potential impairment or damage to the subject's eyes (e.g., hemorrhage, retinal detachment, central corneal ulcer or damage to the optic nerve).
- A congenital anomaly/birth defect.

Important medical events that may not result in death, are not life-threatening, or do not require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

#### 17.2 Visual Acuity (Early Treatment Diabetic Retinopathy Study)

| The logarithm of the minimum angle of resolution ( | |
|---|---|
| | A subject listing of visual acuity will also be produced |



# 17.3 Slit-Lamp Biomicroscopy

| A slit-lamp biomicroscopy |
|---|
| A subject listing of the slit-lamp biomicroscopy parameters will also be |
| produced. |
| 17.4 Dilated Fundoscopy Examination |
| An dilated fundoscopy examination |
| A subject listing of the dilated fundoscopy parameters will also be produced. |
| 17.5 Intraocular Pressure (IOP) |
| Subjects' IOP |
| Subjects 10F |
| . A subject listing of IOP will also be produced |
| 18. Changes from Protocol-Stated Analyses |
| There are no changes from protocol-stated analyses. |
| 19. References |
| No references cited. |
| 20. Revision History |
| Documentation of revision to the SAP will commence after approval of the final version 1.0. |
| 20.1 Revision 01 |
| This revision was issued following |





### 21. Tables

Tables (10 tables) in **boldface** font will be delivered in topline package.

| Table Number | Title | Population |
|---|---|---|
| | Subject Disposition | All Screened |
| Table 14.1.1 | | Subjects |
| Table 14.1.2.1 | Demographics | ITT Population |
| Table 14.1.2.2 | Demographics | Safety Population |
| Table 14.1.2.3 | Participation in Previous Reproxalap Trials | ITT Population |
| Table 14.1.3.1 | Baseline Disease Characteristics | ITT Population |
| Table 14.1.3.2 | Baseline Disease Characteristics | Safety Population |
| Table 14.1.4.1 | Ocular Medical History | ITT Population |



| Table 14.1.4.2 | Non-Ocular Medical History | ITT Population |
|---|---|---|
| Table 14.1.5.1 | Ocular Concomitant Medications | ITT Population |
| Table 14.1.5.2 | Non-Ocular Concomitant Medications | ITT Population |
| Table 14.1.5.3 | Ocular Concomitant Procedures | ITT Population |
| Table 14.1.5.4 | Non-Ocular Concomitant Procedures | ITT Population |
| | Overall Mean Change from Baseline of | ITT Population with |
| | Conjunctival Redness (Ora Calibra Scale) during | Observed Data Only |
| Table 14.2.1.1 | | |
| | Overall Mean Change from Baseline of Conjunctival | PP Population with |
| Table 14.2.1.2 | Redness (Ora Calibra Scale) | Observed Data Only |
| | Overall Mean Change from Baseline of Conjunctival | ITT Population with |
| | Conjunctival Redness (Ora Calibra Scale) | Observed Data Only |
| Table 14.2.1.3 | | |
| | Overall Mean Change from Baseline of Conjunctival | ITT Population with |
| | Conjunctival Redness (Ora Calibra Scale) | Observed Data Only |
| Table 14.2.1.4 | | |
| | Overall Mean Change from Baseline of Conjunctival | ITT Population with |
| Table 14.2.1.5 | Redness (Ora Calibra Scale) | PMM |
| | Overall Mean Change from Baseline of Conjunctival | ITT Population with |
| Table 14.2.1.6 | Redness (Ora Calibra Scale) | MCMC |
| | Overall Mean Change from Baseline of Eye | ITT Population with |
| | Dryness (Visual Analog Scale) | Observed Data Only |
| Table 14.2.2.1 | | |
| | Overall Mean Change from Baseline of Eye | ITT Population with |
| | Dryness (Visual Analog Scale) | Observed Data Only |
| Table 14.2.2.2 | | |
| | Overall Mean Change from Baseline of Ocular | ITT Population with |
| | Discomfort Scale (Ora Calibra Scale) | Observed Data Only |
| Table 14.2.2.3 | | |
| | Overall Mean Change from Baseline of Ocular | ITT Population with |
| | Discomfort Scale (Ora Calibra Scale) | Observed Data Only |
| Table 14.2.2.4 | | |



| T-1-1-44005 | Unanethetized Schirmer's Test | ITT Population with |
|---|---|---|
| Table 14.2.2.5 | | Observed Data Only |
| | Eye Dryness (Visual Analog Scale) | ITT Population with |
| Table 14.2.3.1 | | Observed Data Only |
| | Ocular Discomfort Scale (Ora Calibra Scale) | ITT Population with |
| Table 14.2.3.2 | | Observed Data Only |
| | Ocular Discomfort & Four-Symptom Questionnaire | ITT Population with |
| | (Ora Calibra Scale) | Observed Data Only |
| Table 14.2.3.3 | | |
| | Ocular Discomfort & Four-Symptom Questionnaire | ITT Population with |
| | (Ora Calibra Scale) | Observed Data Only |
| Table 14.2.3.4 | | |
| | Conjunctival Allergen Challenge Ocular Itching Scale | ITT Population with |
| | (Ora Calibra Scale) | Observed Data Only |
| Table 14.2.3.5 | | |
| | Conjunctival Allergen Challenge Ocular Itching Scale | ITT Population with |
| | (Ora Calibra Scale) | Observed Data Only |
| Table 14.2.3.6 | | |
| | Tear Reactive Aldehyde Species | ITT Population with |
| Table 14.2.3.7 | | Observed Data Only |
| | Conjunctival Redness (Ora Calibra Scale) | ITT Population with |
| Table 14.2.3.8 | | Observed Data Only |
| | Conjunctival Redness (Ora Calibra Scale) | ITT Population with |
| Table 14.2.3.9 | | Observed Data Only |
| | Eye Dryness (Visual Analog Scale) | ITT Population with |
| Table 14.2.3.10 | | Observed Data Only |
| | Ocular Discomfort Scale (Ora Calibra Scale) | ITT Population with |
| Table 14.2.3.11 | | Observed Data Only |
| | Overall Mean Change from Baseline of Conjunctival | Initial Cohort |
| | Redness (Ora Calibra Scale) | Population with |
| Table 14.2.4.1 | | Observed Data Only |



| | Overall Mean Change from Baseline of Eye Dryness | Initial | Cohort |
|---|---|---|---|
| | (Visual Analog Scale) | Population | with |
| Table 14.2.4.2 | | Observed Data Only | |
| | Overall Mean Change from Baseline of Eye Dryness | Initial | Cohort |
| | (Visual Analog Scale) | Population | with |
| Table 14.2.4.3 | | Observed Data Only | |
| | Overall Mean Change from Baseline of Ocular | Initial | Cohort |
| | Discomfort Scale (Ora Calibra Scale) | Population | with |
| Table 14.2.4.4 | | Observed Da | ta Only |
| | Overall Mean Change from Baseline of Ocular | Initial | Cohort |
| | Discomfort Scale (Ora Calibra Scale) | Population | with |
| Table 14.2.4.5 | | Observed Da | ta Only |
| | Unanesthetized Schirmer's Test | Initial | Cohort |
| | | Population | with |
| Table 14.2.4.6 | | Observed Da | ta Only |
| | Eye Dryness (Visual Analog Scale) | Initial | Cohort |
| | | Population | with |
| Table 14.2.4.7 | | Observed Data Only | |
| | Ocular Discomfort Scale (Ora Calibra Scale) | Initial | Cohort |
| | | Population | with |
| Table 14.2.4.8 | | Observed Data Only | |
| | Ocular Discomfort & Four-Symptom Questionnaire | Initial | Cohort |
| | (Ora Calibra Scale) | Population | with |
| Table 14.2.4.9 | | Observed Da | ta Only |
| | Tear Reactive Aldehyde Species | Initial | Cohort |
| | | Population | with |
| Table 14.2.4.10 | | Observed Da | ta Only |
| | Conjunctival Redness (Ora Calibra Scale) | Initial | Cohort |
| | | Population | with |
| Table 14.2.4.11 | | Observed Da | ta Only |
| | Eye Dryness (Visual Analog Scale) | Initial | Cohort |
| | | Population | with |
| Table 14.2.4.12 | | Observed Da | ta Only |



| | Ocular Discomfort Scale (Ora Calibra Scale) | Initial Cohort |
|---|---|---|
| Table 14.2.4.13 | | Population with Observed Data Only |
| Table 14.2.5 | Summary of Efficacy Analyses | Multiple Populations |
| Table 14.3.1.1 | Overall Summary of Adverse Events by Treatment Arm | Safety Population |
| Table 14.3.2.1 | Ocular Adverse Events by System Organ Class and Preferred Term | Safety Population |
| Table 14.3.2.2 | Non-Ocular Adverse Events by System Organ Class and Preferred Term | Safety Population |
| Table 14.3.3.1 | Ocular Treatment-Emergent Adverse Events by<br>System Organ Class and Preferred Term | Safety Population |
| Table 14.3.3.2 | Non-Ocular Treatment-Emergent Adverse Events by<br>System Organ Class and Preferred Term | Safety Population |
| Table 14.3.4 | Instillation Site Ocular TEAEs by SOC, PT, and Duration of Time | Safety Population |
| Table 14.3.5.1 | Ocular Treatment-Emergent Adverse Events by<br>System Organ Class, Preferred Term, and Maximal<br>Severity | Safety Population |
| Table 14.3.5.2 | Non-Ocular Treatment-Emergent Adverse Events by<br>System Organ Class, Preferred Term, and Maximal<br>Severity | Safety Population |
| Table 14.3.6.1 | Ocular Treatment-Emergent Adverse Events by<br>System Organ Class, Preferred Term, and Strongest<br>Relationship to Study Procedure | Safety Population |
| Table 14.3.6.2 | Non-Ocular Treatment-Emergent Adverse Events by<br>System Organ Class, Preferred Term, and Strongest<br>Relationship to Study Procedure | Safety Population |
| Table 14.3.7.1 | Ocular Treatment-Emergent Adverse Events by<br>System Organ Class, Preferred Term, Maximal<br>Severity, and Strongest Relationship to Study<br>Procedure | Safety Population |
| Table 14.3.7.2 | Non-Ocular Treatment-Emergent Adverse Events by<br>System Organ Class, Preferred Term, Maximal | Safety Population |



| | Severity, and Strongest Relationship to Study Procedure | |
|---|---|---|
| | Treatment-Emergent Adverse Events That Led to | Safety Population |
| Table 14.3.8 | Premature Discontinuation | |
| Table 14.3.9 | Treatment-Emergent Serious Adverse Events | Safety Population |
| Table 14.3.10 | Visual Acuity (ETDRS) | Safety Population |
| Table 14.3.11.1 | Slit Lamp Biomicroscopy | Safety Population |
| Table 14.3.11.2 | Shift in Slit Lamp Biomicroscopy | Safety Population |
| Table 14.3.12 | Intraocular Pressure | Safety Population |
| Table 14.3.13.1 | Dilated Fundoscopy | Safety Population |
| Table 14.3.13.2 | Shift in Dilated Fundoscopy | Safety Population |
| Table 14.3.14 | Compliance to Study Drug | Safety Population |
| Table 14.3.15 | Exposure to Study Drug | Safety Population |

### 22. Listings

| Listing Number | Title | Population |
|---|---|---|
| | Randomization Schedule | All Randomized |
| Listing 16.1.7 | | Subjects |
| | Subject Disposition | All Randomized |
| Listing 16.2.1.1 | | Subjects |
| Listing 16.2.1.2 | Inclusion/Exclusion and Screen Failure | All Screened Subjects |
| Listing 16.2.2 | Protocol Deviations | All Screened Subjects |
| | Study Population Inclusion | All Randomized |
| Listing 16.2.3.1 | | Subjects |
| Listing 16.2.3.2 | Subjects Affected by COVID-19 | All Screened Subjects |
| Listing 16.2.4.1 | Demographics | All Screened Subjects |
| | Ocular Medical History | All Randomized |
| Listing 16.2.4.2 | | Subjects |
| | Non-Ocular Medical History | All Randomized |
| Listing 16.2.4.3 | | Subjects |



| | Ocular Concomitant Medications | All Randomized |
|---|---|---|
| Listing 16.2.4.4 | | Subjects |
| | Non-Ocular Concomitant Medications | All Randomized |
| Listing 16.2.4.5 | | Subjects |
| Listing 16.2.5.1 | Run-In Instillation | All Screened Subjects |
| | Study Drug Assignment, Instillation, and Replacement | All Randomized |
| Listing 16.2.5.2 | | Subjects |
| | Study Drug Exposure and Dosing Compliance | All Randomized |
| Listing 16.2.5.3 | | Subjects |
| | Study Drug Accountability | All Randomized |
| Listing 16.2.5.4 | | Subjects |
| | Conjunctival Redness (Ora Calibra Scale) | All Randomized |
| Listing 16.2.6.1 | | Subjects |
| | Conjunctival Redness (Ora Calibra Scale) | All Randomized |
| Listing 16.2.6.2 | | Subjects |
| | Eye Dryness (Visual Analog Scale) | All Randomized |
| Listing 16.2.6.3 | | Subjects |
| 10004 | Eye Dryness (Visual Analog Scale) | All Randomized |
| Listing 16.2.6.4 | | Subjects |
| Listing 40.0.5 | Ocular Discomfort Scale (Ora Calibra Scale) | All Randomized |
| Listing 16.2.6.5 | | Subjects |
| Listing 40.0.0 | Ocular Discomfort Scale (Ora Calibra Scale) | All Randomized |
| Listing 16.2.6.6 | | Subjects |
| Linting 46.0.6.7 | Ocular Discomfort & 4-Symptom Questionnaire (Ora | All Randomized |
| Listing 16.2.6.7 | Calibra Scale) | Subjects |
| Linting 46.0.6.0 | Conjunctival Allergen Challenge Ocular Itching Scale | All Randomized |
| Listing 16.2.6.8 | (Ora Calibra Scale) | Subjects |
| Listing 16.2.6.0 | Tear Reactive Aldehyde Species | All Randomized |
| Listing 16.2.6.9 | | Subjects |
| Listing 16.2.6.10 | Unanesthetized Schirmer's Test | All Randomized |
| Listing 16.2.6.10 | | Subjects |
| Listing 16.2.6.11 | Fluorescein Corneal and Conjunctival Staining (Ora | All Randomized |
| Listing 16.2.6.11 | Calibra Scale) | Subjects |



| Listing 16.2.7.1 | All Adverse Events | All Screened Subjects | |
|---|---|---|---|
| Listing 16.2.7.2 | Ocular Adverse Events | All Scree | All Screened Subjects |
| Listing 16.2.7.3 | Non-Ocular Adverse Events | All Scree | ened Subjects |
| Listing 16.2.7.4 | Serious Adverse Events | All Scree | ened Subjects |
| | Visual Acuity | All | Randomized |
| Listing 16.2.8.1 | | Subjects | <b>i</b> |
| | Slit-Lamp Biomicroscopy | All | Randomized |
| Listing 16.2.8.2 | | Subjects | <b>i</b> |
| | Intraocular Pressure (IOP) | All | Randomized |
| Listing 16.2.8.3 | | Subjects | <b>i</b> |
| | Dilated Fundoscopy | All | Randomized |
| Listing 16.2.8.4 | | Subjects | i |
| | Pregnancy Test | All Fem | ale Screened |
| Listing 16.2.8.5 | | Subjects | i. |
| | Tear Collection | All | Randomized |
| Listing 16.2.8.6 | | Subjects | • |